CLINICAL TRIAL: NCT06514911
Title: Primary Closure Versus T-tube Drainage Following Laparoscopic Cholodochotomy in Management of CBD Stones
Brief Title: Laparoscopic Cholodochotomy in Management of CBD Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Khalaf Mohamed, Resident, Department of General Surgery, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-06-25MS
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-06

CONDITIONS: Management of CBD Stones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary closure following Laparoscopic cholodochotomy in management of CBD stones (Active Comparator)
  Interventions: Procedure: primary closure following Laparoscopic cholodochotomy in management of CBD stones
- T-tube drainage following Laparoscopic cholodochotomy in management of CBD stones (Active Comparator)
  Interventions: Procedure: T-tube drainage following Laparoscopic cholodochotomy in management of CBD stones

INTERVENTIONS:
Procedure: primary closure following Laparoscopic cholodochotomy in management of CBD stones — primary closure of cholodochotomy incision in laparoscopic CBD exploration avoiding T-tube insertion
  Arms: primary closure following Laparoscopic cholodochotomy in management of CBD stones
Procedure: T-tube drainage following Laparoscopic cholodochotomy in management of CBD stones — drainage of bile by T-tube insertion in laparpscopic CBD exploration
  Arms: T-tube drainage following Laparoscopic cholodochotomy in management of CBD stones

SUMMARY:
The aim of this study is to compare the outcomes of primary closure of cholodochotomy incision versus T-tube drainage in laparoscopic common bile duct exploration for management of CBD stones and provide evidence-based guidance to the selection of the most appropriate operative technique.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a definitive preoperative diagnosed with CBD stones.
2. a CBD diameter of ≥1 cm.
3. patients are fit for surgery

Exclusion Criteria:

1. patients with liver cirrhosis.
2. a CBD diameter of <1 cm
3. malignancy in the biliary tract or CBD stricture .
4. patients are not fit for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
biliary leakage in the management of CBD stones | 3 days after the operation
  peritoneal collection of bile after common bile duct exploration

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Cianci P, Restini E. Management of cholelithiasis with choledocholithiasis: Endoscopic and surgical approaches. World J Gastroenterol. 2021 Jul 28;27(28):4536-4554. doi: 10.3748/wjg.v27.i28.4536. PMID 34366622
- [Background] Tan D, Zhang Y. Differences in Outcome and Comparison of Stress and Immune Status in Patients with Recurrent Common Bile Duct Stones after Biliary Tract Surgery Choosing Three Procedures (ERCP, OCBDE, and LCBDE) for Treatment. Comput Math Methods Med. 2022 Jan 5;2022:9197990. doi: 10.1155/2022/9197990. eCollection 2022. PMID 35035527
- [Background] Hua J, Lin S, Qian D, He Z, Zhang T, Song Z. Primary closure and rate of bile leak following laparoscopic common bile duct exploration via choledochotomy. Dig Surg. 2015;32(1):1-8. doi: 10.1159/000368326. Epub 2015 Jan 22. PMID 25613528